CLINICAL TRIAL: NCT01105598
Title: A Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ETC-1002 in Subjects With Mild Dyslipidemia
Brief Title: A Multiple Ascending Dose Study of ETC-1002 in Subjects With Mild Dyslipidemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETC-1002-002
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Mild Dyslipidemia
MeSH Terms: interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Subjects (6 active/2 placebo) with mild dyslipidemia in Phase 1 Unit
  Interventions: Drug: ETC-1002 or placebo
- Cohort 2 (Experimental): Subjects (6 active/2 placebo) with mild dyslipidemia in Phase 1 Unit
  Interventions: Drug: ETC-1002 or placebo
- Cohort 3 (Experimental): Subjects (6 active/2 placebo) with mild dyslipidemia in Phase 1 Unit
  Interventions: Drug: ETC-1002 or placebo
- Cohort 4 (Experimental): Subjects (6 active/2 placebo) with mild dyslipidemia in Phase 1 Unit
  Interventions: Drug: ETC-1002 or placebo
- Cohort 5 (Experimental): Free-living subjects (18 active/6 placebo) with mild dyslipidemia
  Interventions: Drug: ETC-1002 or placebo

INTERVENTIONS:
Drug: ETC-1002 or placebo — ETC-1002 (ascending dose), daily for 14 days
  Arms: Cohort 2; Cohort 3; Cohort 4
Drug: ETC-1002 or placebo — ETC-1002 (optimized dose), daily for 28 days
  Arms: Cohort 5
Drug: ETC-1002 or placebo — ETC-1002 (20 mg), daily for 14 days
  Arms: Cohort 1

SUMMARY:
This Phase 1, double-blind (sponsor open) study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of ETC-1002 given to subjects with mild dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects of non-child bearing potential as determined by medical history, physical examination, vital signs, ECG, and clinical laboratory measurements
* Fasting low density lipoprotein-cholesterol (LDL-C) of 100-160 mg/dL
* Fasting triglycerides (TG) of 100-350 mg/dL (Cohort 5 only)
* Body Mass Index (BMI) of 18-32 kg/m2 (Cohort 1 to 4 only) or 18-36 (Cohort 5 only) and body weight >50 kg

Exclusion Criteria:

* Clinically significant disease that requires a physician's care and/or would interfere with study evaluations
* Alanine aminotransferase (ALT) or aspartate amino transferase (AST) >1.2 x ULN; serum creatinine >ULN; hemoglobin <12.0 g/dL; other clinical lab tests (with the exception of ALT, AST, serum creatinine and hemoglobin) outside normal or protocol specified limits that are determined by the Investigator to be clinically significant
* Use of tobacco or tobacco products
* Use of any prescription or nonprescription drugs, vitamins, or dietary supplements within 14 days prior to randomization with the exception of lipid regulating drugs or supplements containing niacin >500 mg/day or fish oil which will not have been used for 3 months prior to randomization
* Other exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2010-04-20 (Actual); Primary Completion 2010-10-02 (Actual); Study Completion 2010-10-02 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability using adverse event reports, physical exams, vitals signs, ECGs, and clinical lab values | 14 or 28 days

SECONDARY OUTCOMES:
Characterization of pharmacokinetic parameters and percent change from baseline in pharmacodynamic endpoints | 14 or 28 days
  Pharmacodynamic endpoints include total cholesterol, low density lipoprotein-cholesterol (LDL-C), triglycerides (TG), high density lipoprotein-cholesterol (HDL-C) and free fatty acids (FFA)

CONTACTS AND LOCATIONS:
Overall Officials: Jim C Khalifa, MD, Study Director — Esperion Therapeutics, Inc.
Locations (1):
- Jasper Clinic, Inc., Kalamazoo, Michigan, United States